CLINICAL TRIAL: NCT00622674
Title: Phase I Study of Bortezomib (Velcade) and Cetuximab (Erbitux) for Patients With Solid Tumors Expressing EGFR
Brief Title: Bortezomib and Cetuximab in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000586671; UMN-2005LS037 (Other: CPRC, University of Minnesota); MILLENNIUM-X05160 (Other: Millennium Pharm Inc.); UMN-0506M7030372 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2008-02-22; First posted 2008-02-25 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2010-04

CONDITIONS: Breast Cancer; Colorectal Cancer; Head and Neck Cancer; Kidney Cancer; Lung Cancer; Pancreatic Cancer; Sarcoma; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: recurrent breast cancer; recurrent non-small cell lung cancer; recurrent small cell lung cancer; recurrent colon cancer; recurrent pancreatic cancer; recurrent head and neck cancer; recurrent sarcoma; recurrent kidney cancer; recurrent renal cell cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Head and Neck Neoplasms; Kidney Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Sarcoma; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Colonic Neoplasms; Carcinoma, Renal Cell | interventions — Cetuximab; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib and Cetuximab (Experimental): The starting dose of bortezomib will be 1.3 mg/m2 with a 0.1 increment increase with each successive dose level to a maximum of 2.0 mg/m2. A loading dose of cetuximab will be given on day 1 (400 mg/m2) followed by a weekly dose of 250 mg/m2.
  Interventions: Biological: cetuximab; Drug: bortezomib

INTERVENTIONS:
Biological: cetuximab — A loading dose of cetuximab will be given on day 1 (400 mg/m2) followed by a weekly dose of 250 mg/m2.
  Other Names: Erbitux
Drug: bortezomib — The starting dose of bortezomib will be 1.3 mg/m2 with a 0.1 increment increase with each successive dose level to a maximum of 2.0 mg/m2.
  Other Names: Velcade

SUMMARY:
RATIONALE: Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving bortezomib together with cetuximab may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of bortezomib when given together with cetuximab in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose of bortezomib when given together with cetuximab in patients with advanced solid tumors expressing epidermal growth factor receptor (EGFR).

Secondary

* To obtain preliminary information about the anti-tumor activity of bortezomib and cetuximab.

OUTLINE: This is a dose-escalation study of bortezomib.

Patients receive bortezomib intravenously (IV) on days 1 and 8 and cetuximab IV over 60-90 minutes on days 1, 8, and 15. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After the maximum tolerated dose (MTD) is determined, an additional 10 patients are treated at the MTD.

After completion of study treatment, patients are followed periodically for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of solid tumor that overexpresses epidermal growth factor receptor (EGFR) including, but not limited to, the following:

  * Breast cancer
  * Lung cancer
  * Colon cancer
  * Pancreatic cancer
  * Head and neck cancer
  * Kidney cancer
  * Sarcoma
* Advanced disease

  * Must have failed or become intolerant to prior standard therapy and is no longer likely to respond to such therapy
* Measurable or nonmeasurable disease
* ECOG performance status 0-1
* ANC ≥ 1,500/mm³
* Platelet count > 100,000/mm³
* Hemoglobin > 9 g/dL
* Bilirubin < 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase < 3.0 times ULN (5.0 times ULN if liver has tumor involvement)
* Aspartate aminotransferase (AST) and alanine aminotransferase (*ALT) < 3.0 times upper limit of normal (ULN) (5.0 times ULN if liver has tumor involvement)
* Creatinine clearance > 30 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* Recovered from all prior therapy
* Prior systemic chemotherapy, immunotherapy, or biological therapy allowed
* At least 14 days since prior radiotherapy or systemic therapy
* At least 30 days since prior investigational agents
* At least 14 days since other prior investigational drugs (for reasons other than the treatment of cancer)

Exclusion Criteria:

* Untreated or symptomatic central nervous system (CNS) metastases
* Concurrent serious systemic disorders (e.g., active infection) that, in the opinion of the investigator, would compromise the safety of the patient or compromise the patient's ability to complete the study
* Uncontrolled diabetes
* Myocardial infarction within the past 6 months
* New York Heart Association (NYHA) class III or IV heart failure
* Uncontrolled angina
* Severe uncontrolled ventricular arrhythmias
* Evidence of acute ischemia or active conduction system abnormalities by ECG
* Peripheral neuropathy Common Terminology Criteria for Adverse Events (CTCAE) grade > 2
* Known hypersensitivity to bortezomib, boron, or mannitol
* Serious medical or psychiatric illness likely to interfere with study participation
* Prior bortezomib and/or cetuximab
* Concurrent filgrastim (G-CSF) or other hematologic support during course 1 of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2005-11; Primary Completion 2009-08 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of bortezomib | At end of Cycle 1 (Week 3)
  The standard Phase I design will be used to determine the maximum tolerated dose of bortezomib when given with weekly cetuximab. The MTD is defined as the highest dose studied for which the incidence of dose limiting toxicity (DLT) was less than 33%.

SECONDARY OUTCOMES:
Disease response as measured by RECIST criteria | At Week 4
  The best overall response is the best response recorded from registration until disease progression/recurrence, taking as reference for progressive disease the smallest measurements recorded since registration.

CONTACTS AND LOCATIONS:
Overall Officials: Arkadiusz Dudek, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States